CLINICAL TRIAL: NCT01864161
Title: Endovenous Versus Liposomal Iron in CKD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIANCA79
Record Dates: First submitted 2013-05-24; First posted 2013-05-29 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2013-01

CONDITIONS: Iron Deficiency Anemia; Chronic Kidney Disease
MeSH Terms: conditions — Anemia, Iron-Deficiency; Renal Insufficiency, Chronic | interventions — ferlixit

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- oral liposomal iron (Experimental): patients receive a dose of liposomal 30 mg/die iron (equivalent to 1 cp Sideral forte).
  Interventions: Drug: Liposomal iron
- endovenous iron (Active Comparator): patients receive a total dose 1000 mg of intravenous iron gluconate divided into administrations of 125 mg diluted in 250 mL normal saline infused weekly for 3 months
  Interventions: Drug: gluconate iron

INTERVENTIONS:
Drug: gluconate iron — FERLIXIT fl 15mg/kg divided into weekly administrations of 125mg up to a maximum of 1000mg
  Other Names: FERLIXIT
  Arms: endovenous iron
Drug: Liposomal iron — Sideral forte 30 mg/die
  Other Names: Sideral forte
  Arms: oral liposomal iron

SUMMARY:
Anemia is a common complication in patients with chronic kidney disease (CKD). In addition to erythropoietin deficiency, many studies have identified iron deficiency as a cause of anemia in CKD patients. Most patients with CKD are iron deficient because of: inadequate intake and absorption, gastroenteric bleeding, urinary iron loss in patient with significant proteinuria. The iron treatment is pivotal to manage anemic patients with CKD: the prescription of iron is usually oral because of practicality and safety, but often it is inevitable to administer intravenous iron because of gastroenteric malabsorption, intolerance to oral administration, irregular intake. There're few randomized controlled studies about the efficacy of oral iron versus intravenous iron in patients not on dialysis; most of them demonstrate superiority of intravenous therapy to restore iron deficiency and hemoglobin levels. A particular formulation of iron, liposomal iron has a high gastroenteric absorption and high bioavailability with lower incidence of side effects. The investigators study aims to evaluate the efficacy of treatment with liposomal oral iron compared to intravenous iron in CKD anemic patients not on dialysis in the presence of iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Signed written informed consent;
* Glomerular filtration rate (GFR) ≤ 60 mL/min (MDRD GFR calculated according to 4 variables);
* hemoglobin ≤ 12g/dL;
* Ferritin ≤ 100ng/mL with transferrin saturation (TSAT) ≤ 25%;
* If erythropoiesis stimulating agents (ESA) therapy, stable dose for at least three months;

Exclusion Criteria:

* Infectious diseases;
* bleeding in the preceding six months;
* History of malignancy tumor in the last 3 years;
* Anemia case different from that resulting from CKD;
* vitamin B12 and folate deficiency;
* Surgery of any kind in the last three months;
* systemic haematological disease;
* Blood Transfusions, therapy with intravenous or oral iron in the last three months;
* Severe liver disease / test positive for hepatitis C virus (HCV) and hepatitis B virus (HBV);
* Abuse of alcohol and drugs in the preceding six months;
* immunosuppressive therapy ;
* Significant weight loss;
* Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
modification in hemoglobin levels | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Federico II University, Naples, Naples, Italy